CLINICAL TRIAL: NCT00206115
Title: A 6-week, Multicenter, Double-blind, Double-dummy, Randomized Comparison of the Efficacy & Safety of Sustained-Release Formulation Quetiapine Fumarate (SEROQUEL) & Placebo in the Treatment of Acutely Ill Patients With Schizophrenia
Brief Title: SR-Registration Study 1, ROW: Efficacy and Safety of Seroquel® in the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1444C00132
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenic Disorder
Keywords: Schizophrenic disorder
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Seroquel Sustained Release (SR)
Drug: Seroquel Immediate Release (IR)
Drug: Placebo

SUMMARY:
The purpose of this 6-week study is to determine whether treatment with Seroquel® Sustained Release (SR) is more effective than placebo in the treatment of acute schizophrenia.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* To be considered for this study the patients should be aged between 18 to 65 years, need to suffer from schizophrenia and must be willing to participate.

Exclusion Criteria:

* Patients that suffer from psychiatric disorders other than schizophrenia including drug abuse and dependence, or medical conditions such as specific kidney, heart or thyroid problems, and patients with a known lack of response to drugs for schizophrenia will not be considered for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535
Dates: Start 2004-11; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be the change from baseline of the Positive and Negative Syndrome Scale (PANSS) total score at the end of treatment at Day 42.

SECONDARY OUTCOMES:
Efficacy
To demonstrate a higher PANSS response rate
To demonstrate superior Clinical Global Impressions (CGI) response

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca CNS Medical Science Director, MD, Study Director — AstraZeneca
Locations (31):
- Bulgaria (4):
  - Research Site, Burgas
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Sofia- Novi Iskar
- Greece (4):
  - Research Site, Athens
  - Research Site, Chania
  - Research Site, Corfu
  - Research Site, Thessaloniki
- India (4):
  - Research Site, Chennai
  - Research Site, Karnataka
  - Research Site, Lucknow
  - Research Site, New Delhi
- Indonesia (3):
  - Research Site, Jakarta, DKI Jakarta
  - Research Site, Bandung, West Java
  - Research Site, Surabaya
- Philippines (5):
  - Research Site, Cebu
  - Research Site, Davao City
  - Research Site, Mandaluyong
  - Research Site, Manila
  - Research Site, Pasig
- Romania (2):
  - Research Site, Brasov
  - Research Site, Bucharest
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Africa (7):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Medunsa, Pretoria
  - Research Site, Bloemfontein
  - Research Site, Ga-Rankuwa
  - Research Site, Johannesburg
  - Research Site, Lyttelton Manor
  - Research Site, Pretoria

REFERENCES:
- [Derived] Kahn RS, Schulz SC, Palazov VD, Reyes EB, Brecher M, Svensson O, Andersson HM, Meulien D; Study 132 Investigators. Efficacy and tolerability of once-daily extended release quetiapine fumarate in acute schizophrenia: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2007 Jun;68(6):832-42. doi: 10.4088/jcp.v68n0603. PMID 17592906